CLINICAL TRIAL: NCT00646854
Title: A Randomized Phase III Study to Evaluate the Efficacy of Chemoimmunotherapy With the Monoclonal Antibody Campath-1H (Alemtuzumab) Given in Combination With 2-weekly CHOP Versus 2-weekly CHOP Alone and Consolidated by Autologous Stem Cell Transplant, in Young Patients With Previously Untreated Systemic Peripheral T-cell Lymphomas
Brief Title: Alemtuzumab and CHOP in T-cell Lymphoma
Acronym: ACT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: GCP-unit at Aarhus University Hospital, Aarhus, Denmark (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-006130-17
Record Dates: First submitted 2008-02-14; First posted 2008-03-31 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: Lymphoma, T-Cell; Lymphoma, T-Cell, Peripheral; MabCampath; Campath; CHOP-14; CD52 expression
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Active Comparator)
  Interventions: Drug: CHOP14 chemotherapy (see specification under Arm B) plus G-CSF
- Arm B (Experimental)
  Interventions: Drug: CHOP14 chemotherapy (cyclophosphamide, hydroxydaunorubicin, vincristin, prednison) plus G-CSF, combined with alemtuzumab

INTERVENTIONS:
Drug: CHOP14 chemotherapy (cyclophosphamide, hydroxydaunorubicin, vincristin, prednison) plus G-CSF, combined with alemtuzumab — Cyclophosphamide 750 mg/m2 i.v. on day 1 Hydroxydaunorubicin 50 mg/m2 i.v. on day 1 Vincristin 1 mg/m2 i.v. day 1 (max. 2mg) Prednisone 50 mg/m2 p.o. day 1 to 5 Alemtuzumab 30 mg s.c.on day 1 of CHOP-14 cycles 1-4
  Arms: Arm B
Drug: CHOP14 chemotherapy (see specification under Arm B) plus G-CSF — 6 cycles of CHOP every 2 weeks
  Arms: Arm A

SUMMARY:
The purpose of this study is to determine efficacy and safety of the monoclonal antibody MabCampath® (alemtuzumab) combined with chemotherapy in the treatment of T-cell lymphoma.

DETAILED DESCRIPTION:
First International phase III T-cell lymphoma study Indication:Newly diagnosed non-cutaneous peripheral T-cell lymphoma Study objectives:Determination of the efficacy and safety of the monoclonal antibody MabCampath® (alemtuzumab) combined with two-weekly CHOP supported by G-CSF Primary Endpoint: Event-Free-Survival (EFS) Study Design: International open-label, multicentre, randomized Phase III Study

Study Medication: Patients are randomized to six cycles of two-weekly CHOP plus G-CSF with or without alemtuzumab given subcutaneously 30 mg day 1 in combination with chemotherapy cycles 1-4. Patients in CR, CRu and PR after the 6 cycles of CHOP14 combined or not with alemtuzumab will receive a consolidation with high-dose chemotherapy followed by autologous stem cell transplantation.

Patient Population: Patients > 18 yrs with newly diagnosed non-cutaneous, non-leukemic PTCL, except alk-protein positive and negative anaplastic large cell lymphoma Planned Sample Size: 308 young patients (18-60 yrs) registered and randomized Total Number of Centers: This study will be proposed to main European and Australian Study Groups.

ELIGIBILITY:
Inclusion criteria:

* Previously untreated patients with newly diagnosed peripheral T-cell lymphoma of stage I bulk (≥ 7.5 cm) and stages II to IV.
* Patients with a confirmed histologic diagnosis of peripheral T-cell NHL according to the WHO classification:
* Peripheral T-cell lymphoma, unspecified (PTCL NOS)
* Angioimmunoblastic T-cell lymphoma
* Enteropathy-type T cell lymphoma
* Subcutaneous panniculitis-like T-NHL (gamma-delta T-cell lymphoma)
* Hepatosplenic T-cell lymphoma
* Extranodal NK/T cell lymphoma, nasal type
* Age 18-60 years at time of randomization
* Life expectancy of 3 months or longer
* ECOG performance status (PS) 0, 1 or 2 at the time of randomization. However, PS 3 will be acceptable if lymphoma-related.
* Measurable disease (defined as at least one lesion with two measurable perpendicular diameters of which at least one should be >= 15 mm).
* Written informed consent

Exclusion Criteria:

* Patients with NK/T-NHL of the following type:
* Precursor T cell lymphoblastic lymphoma/leukemia
* All mature T cell leukemias (T-PLL, ATLL, NK cell leukemia, T-LGL, HTLV1-pos ATL)
* Alk-positive and negative anaplastic large cell lymphoma
* Blastic NK cell lymphoma
* Cutaneous T-cell lymphoma, transformed or not
* Concurrent severe and/or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection), which could compromise participation in the study.
* Known hypersensitivity to murine or chimeric antibodies or proteins
* Severe cardiac dysfunction (NYHA classification II-IV, Appendix H) or LVEF < 45 %
* Significant renal dysfunction, i.e. serum creatinin >2 times upper normal level (UNL), unless related to NHL
* Significant hepatic dysfunction (total bilirubin >2 times UNL or transaminases >= 2.5 times UNL), unless related to NHL
* Impaired pulmonary functions; in this case, the patient is to be excluded if the resultant pulmonary function test shows FEV1<50% or a diffusion capacity <50% of the reference values
* Suspected or documented Central Nervous System involvement by NHL
* Patients known to be HIV-positive
* Patients with active, uncontrolled infections, especially known seropositivity for HCV or HbsAg
* Patients with uncontrolled asthma or allergy, requiring systemic steroid treatment
* Prior treatment with chemotherapy, radiotherapy or immunotherapy for this lymphoma, except local radiotherapy in case of extranodal NK/T cell lymphoma, nasal or nasal type
* History of active cancer during the past 5 years, except basal carcinoma of the skin or stage 0 cervical carcinoma
* Unwillingness or inability to comply with the protocol
* Simultaneous participation in any other study protocol
* Pregnant and nursing women (Women of childbearing potential should use safe anticonceptives) Contraceptive pills, intrauterine devices, injection of prolonged gestagen, subdermal implantation, hormonal vaginal devices and transdermal patches are considered as safe contraceptive methods).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Event-free Survival | The EFS is defined by the time between day of randomization until an event occurs, up to 96 months

SECONDARY OUTCOMES:
Overall survival | From the time of randomisation to date of last follow-up or death, up to 96 months
Overall response rate | from date of randomization to date of primary response assessment, up to 96 months
Overall response rate related to the CD52 expression | From date of randomization to date of primary response assessment, up to 96 months
Tumor control or time-to-progression | time of randomization to last follow-up or time of disease progression, up to 96 months
Safety measured as number of adverse events (AEs) and serious adverse events (SAEs) | from randomization to closure of study, up to 96 months
Feasibility of successful stem cell harvest i.e. >/=2E6 CD34 positive cells | from start of priming regimen to time of assessment of stem cell harvest, up to 96 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco d'Amore, Prof, Principal Investigator — Dept. of Hematology, Århus University Hospital, Denmark
Locations (59):
- Austria (4):
  - AKH Linz, Linz
  - Krankenhaus der Elisabethinen, Linz
  - Center for Clinical Cancer and Immunology Trials, Salzburg
  - Hanusch Krankenhaus, Vienna
- Belgium (12):
  - ZNA Middelheim, Antwerp
  - ZNA Stuivenberg, Antwerp
  - AZ St Jan, Bruges
  - UZ VUB, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Hôpital de Jolimont, Haine-St-Paul
  - UZ Gasthuisberg, Leuven
  - CHR de la Citadelle, Liége
  - Clinique St Pierre, Ottignies
  - Heilig-Hartziekenhuis, Roeselare
  - Clinique de Mont-Godinne, Yvoir
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - University Hospital Kralovske Vinohrady, Prague
  - University Hospital Motol, Prague
- Denmark (6):
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
  - Vejle Hospital, Vejle
- Finland (5):
  - Helsinki University Central Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Tampere University Hospital, Tampere
  - Turku University Central Hospital, Turku
- Germany (3):
  - Charite Universitätsmedizin Berlin, Berlin
  - Krankenhaus Nordwest, Frankfurt
  - University Hospital Regensburg, Regensburg
- Netherlands (13):
  - Meander Medical Center, Amersfoort
  - Vrije University Medical Center, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leids University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - University Medical Center St. Radboud, Nijmegen
  - Erasmus Medical Center - Centrum, Rotterdam
  - Erasmus Medical Center Daniel, Rotterdam
  - Haga Ziekenhuis, loc. Leyenburg, The Hague
  - Isala Klinieken, Sophia, Zwolle
- Norway (4):
  - Radium Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of Nothern Norway, Tromsø
  - St. Olavs Hospital, Trondheim
- Marie Sklodowska-Curie Memorial Institute Cancer Center, Warsaw, Poland
- Portugal (2):
  - IPO Lisboa, Lisbon
  - IPO Porto, Porto
- Sweden (4):
  - Sunderby Hospital, Luleå
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Norrlands University Hospital, Umeå